CLINICAL TRIAL: NCT04924426
Title: Interest of Triphenyl Tetrazolium Chloride (TTC) for the Early Diagnosis of Acute Myocardial Infarction at Autopsy
Brief Title: Interest of TTC for the Early Diagnosis of Acute Myocardial Infarction at Autopsy
Acronym: INFARCTOPSY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0283
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Myocardial Infarction
Keywords: Early Acute Myocardial Infarction; TTC; Sudden death; Early markers; biochemicla markers
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — myocardial fragments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AMI: Patients with AMI
  Interventions: Procedure: TTC immersion
- Patients with no AMI: Patients with no AMI
  Interventions: Procedure: TTC immersion

INTERVENTIONS:
Procedure: TTC immersion — TTC immersion

SUMMARY:
Ischemic heart disease is the leading cause of death worldwide and the leading cause of sudden cardiac death. However, its post-mortem diagnosis is particularly difficult because the gross examination of the heart is usually normal at the autopsy . The diagnosis is therefore often based on a set of indirect arguments, such as the patient's medical and clinical history and the degree of occlusion of the coronary arteries. The formal diagnosis of acute myocardial infarction (AMI) currently relies on standard histological examination. However, histological findings often require a prolonged survival time of several hours to be highlighted. Triphenyltetrazolium chloride (TTC) is a salt that reacts with lactate dehydrogenases contained in still viable myocardial cells, forming a red pigment visible to the naked eye, (1,3,5 triphenylformazan). Ischemia-induced cell death, which occurs within minutes of the causative event, is responsible for the leakage of lactate deshydrogenase into the extracellular medium and thus results in the absence of formazan formation in the infarcted area, which displays an easily identifiable pale unstained color. It has been suggested that the use of TTC would allow the identification of MI as early as one hour of survival in animal models, before the usual macroscopic and microscopic signs are visible. It could therefore represent an attractive forensic tool for the early diagnosis of AMI at the autopsy.

ELIGIBILITY:
Inclusion criteria:

* Adult patients autopsied at the Forensic Institute of the CHU of MONTPELLIER whose ante-mortem (medical history, cardiovascular risk factors, clinical history) and autopsy data (significant coronary stenosis associated or not with an endoluminal thrombus, scars of old infarction, absence of other identified cause of death) suggest AMI as the cause of death.
* Known survival time and postmortem interval.

Exclusion criteria:

- Putrefied bodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspicion of death due to acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Negative colorimetric reaction to TTC of infarcted myocardial tissue | day 1
  Negative colorimetric reaction to TTC of infarcted myocardial tissue

SECONDARY OUTCOMES:
Survival time (time from initial symptoms to death) | day 1
  Survival time (time from initial symptoms to death)
Post-mortem interval (time from death to autopsy) | day 1
  Post-mortem interval (time from death to autopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Antoine Peyron, PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC